CLINICAL TRIAL: NCT01863251
Title: Atomoxetine for ATS and Opioid Dependence During Buprenorphine Maintenance Treatment in Malaysia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202009750
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Opiate Dependence; Stimulant Dependence
Keywords: Opiates; ATS; HIV Risks
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atomoxetine (Experimental): Patients assigned to atomoxetine will receive atomoxetine 40 mg daily, beginning on Day 5. Atomoxetine dose will be increased to 80 mg daily for all patients beginning on Day 12. Atomoxetine will be increased to 120 mg daily for patients with persistent ATS use after 4 weeks of treatment.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Placebo inactive medication
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine
  Other Names: Stratera

SUMMARY:
To evaluate the tolerability, acceptability and potential effect size of the efficacy of 4 months of atomoxetine treatment for patients with co-occurring ATS and heroin dependence (COATS) receiving buprenorphine maintenance treatment (BMT) and educational drug and HIV risk reduction counseling (EDRC).

DETAILED DESCRIPTION:
The Specific Aims of the proposed study are:

1. To evaluate the tolerability, acceptability and potential effect size of the efficacy of 4 months of atomoxetine treatment for patients with co-occurring ATS and heroin dependence (COATS) receiving buprenorphine maintenance treatment (BMT) and educational drug and HIV risk reduction counseling (EDRC).
2. To better characterize patients with co-occurring ATS and heroin dependence (with regard to disturbances of mood, impulse control, executive functioning and patterns of drug use during MMT) and to evaluate the effects of atomoxetine on mood, impulsivity, and executive functioning (including attention, concentration, memory, and decision-making characteristics).
3. To provide training in drug abuse treatment, HIV prevention and treatment, and drug abuse clinical research to drug abuse clinical researchers and clinicians in Kota Bharu, Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Meet Opioid and Amphetamine-type stimulant (ATS)dependence, as assessed by the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM-IV) (SCID) and documented by opioid-positive and ATS positive urine tests.
* Report at least 2 or more days per week of ATS use over the past month.

Exclusion Criteria:

* Hypersensitivity to atomoxetine;
* Current use of a monoamine oxidase inhibitor (MAOI) or use within the preceding 2 weeks;
* Suffer from narrow angle glaucoma; pheochromocytoma; severe cardiovascular disorder; liver enzymes greater than 3 times the upper limit of normal; liver failure or acute hepatitis;
* Pregnancy or breast feeding;
* Current suicide or homicide risk;
* Current psychotic disorder or major depression;
* Inability to understand the protocol or assessment questions.
* A physician reviews the results of all baseline assessments and laboratory and other medical tests (CBC, chemistries, liver enzymes, HIV and Hepatitis B and C, EKG, chest x-ray), takes a medical history, and performs a physical examination in order to confirm the patient's eligibility for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
ATS (Amphetamine-type stimulant) Use | 4 months
  The primary evaluation of the effect size in the proposed study will be based on the overall proportions of urine tests negative for ATS and days per month abstinent from ATS use during the 16 week active study period.

SECONDARY OUTCOMES:
Retention | 4 months
  treatment retention
HIV Risks | 4 months
  Reductions in HIV Risk Behaviors, as assessed by computer-assisted self-report inventory
Functional status | 4 months
  changes in functional outcomes (assessed by the ASI).

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Schottenfled, M.D., Principal Investigator — Yale University; Vicknasingam B Kasinather, Ph.D., Principal Investigator — Univerisiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Malaysia